CLINICAL TRIAL: NCT04436731
Title: Sex Disparities in Hypoxic Sympatholysis and Impact of Obesity
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Principal Investigator, Jacqueline K Limberg, PhD, Assistant Professor, University of Missouri-Columbia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2022525
Record Dates: First submitted 2020-06-08; First posted 2020-06-18 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Obesity; Healthy; Vasoconstriction; Vasodilation
MeSH Terms: conditions — Obesity; Aneurysm | interventions — Phenylephrine; Dexmedetomidine; Phentolamine; Norepinephrine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Hypoxia Exposure (Experimental): A physician will place a catheter in the brachial artery for intra-arterial pharmacological infusions. The following drugs will be administered to each participant under room air (normoxic) and low oxygen (hypoxic) conditions: phenylephrine, dexmedetomidine, norepinephrine, phentolamine (see Interventions for details).
  Interventions: Other: Hypoxia Exposure; Drug: Phenylephrine; Drug: Dexmedetomidine; Drug: Phentolamine; Drug: Norepinephrine

INTERVENTIONS:
Other: Hypoxia Exposure — Systemic oxygen levels will be titrated to attain hypoxemia as assessed by pulse oximetry.
Drug: Phenylephrine — Phenylephrine (0.0625 mcg/dL/min) will be locally infused via brachial artery catheter during the final 3 min of normoxia and hypoxia.
  Other Names: Phenylephrine Hydrochloride
Drug: Dexmedetomidine — Dexmedetomidine (12.5 ng/dL/min) will be locally infused via brachial artery catheter during the final 3 min of normoxia and hypoxia.
Drug: Phentolamine — Phentolamine will be locally infused via brachial artery catheter for 10 min before baseline measurement (12 mcg/dL/min) and the infusion will continue at a maintenance rate (5 mcg/dL/min) during acute normoxia and hypoxia.
  Other Names: Phentolamine mesylate
Drug: Norepinephrine — Regional forearm infusion at 8 ng/dL/min via brachial artery catheter during normoxia and hypoxia exposures

SUMMARY:
Patients with sleep apnea are at increased risk of developing cardiovascular disease - with women at potentially greater risk than men. Contributing mechanisms are not well understood, but may be related to how women respond to low oxygen and, given over 70% of patients with sleep apnea are obese, the impact of obesity. This project seeks to increase our understanding of mechanisms that may contribute to sex differences in the cardiovascular response to low oxygen with the hope that this knowledge will improve the efficacy of current therapies and support the discovery of novel therapeutics.

ELIGIBILITY:
Inclusion Criteria:

* 18-45 years of age (premenopausal)
* Healthy weight (BMI ≥18 and ≤25 kg/m2)
* Obese (BMI ≥30 kg/m2)

Exclusion Criteria:

* Pregnancy, breastfeeding, oral hormonal contraceptive use
* Diagnosed sleep apnea or Oxygen desaturation index >10 events/hr
* Current smoking/Nicotine use
* Increased risk of bleeding, pro-coagulant disorders, clotting disorders, anticoagulation therapy
* Nerve/neurologic disease
* Cardiovascular, hepatic, renal, respiratory disease
* Blood pressure ≥140/90 mmHg
* Diabetes, Polycystic ovarian syndrome
* Communication barriers
* Prescription medications, Sensitivity to lidocaine

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 104 (Estimated)
Dates: Start 2020-12-09 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in forearm vascular conductance with intra-arterial drug infusion | Continuous measurement of vascular conductance during infusion of each drug (final 3 min of normoxia and hypoxia).
  Vascular conductance is an index of vascular tone and is measured using a technique called venous occlusion plethysmography.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Missouri-Columbia, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: No